CLINICAL TRIAL: NCT04711174
Title: Optimization for Laryngeal Mask Removal Strategy and Evaluation of Transitional Criteria From PACU in Children
Status: Completed | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: LMA removal strategy
Record Dates: First submitted 2021-01-04; First posted 2021-01-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-04

CONDITIONS: Complication of Device Removal
Keywords: LMA removal; evaluation of transitional criteria from PACU

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- movement,high Aldrete score group (MH group): LMA removal be conducted when the child's spontaneous respiratory recovers with body movement spontaneously, and the child be transited from PACU when Aldrete score reaches 9
  Interventions: Behavioral: LMA removal
- movement,low Aldrete score group (ML group): LMA removal be conducted when the child's spontaneous respiratory recovers with body movement spontaneously, and the child be transited from PACU when Aldrete score reaches 7
  Interventions: Behavioral: LMA removal
- sedation,high Aldrete score group (SH group): LMA removal be conducted when the child's spontaneous respiratory recovers but with no body movement, and the child be transited from PACU when Aldrete score reaches 9
  Interventions: Behavioral: LMA removal
- sedation,low Aldrete score group (SL group): LMA removal be conducted when the child's spontaneous respiratory recovers but with no body movement, and the child be transited from PACU when Aldrete score reaches 7
  Interventions: Behavioral: LMA removal

INTERVENTIONS:
Behavioral: LMA removal — the timing when conducting LMA removal
  Other Names: Aldrete score

SUMMARY:
Laryngeal mask airway(LMA) is now a widely accepted airway device in general anesthesia for children. LMA removal after operation is always practiced in post-anesthesia-care-unit(PACU). The removal timing depends on recovery of spontaneous respiration and wash-out of inhalation anesthetics. This study focuses on the optimization for LMA removal strategy. Moreover, this study also discusses the transitional criteria from PACU to the ward.

DETAILED DESCRIPTION:
The study recruits 180 children aged under 6-year-old undergoing elective general anesthesia. Laryngeal mask is used in procedure. The children are carried into PACU to get monitored and removal the LMA. The children are randomized into 4 groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged under 6 years old undergoing selected eye surgery
* Scheduled for general anesthesia

Exclusion Criteria:

* With systemic disease
* Respiratory system deformity
* Respiratory infection in 4 weeks

Max Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: children
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
baseline heart rate | before induction
  heart rate before induction
heart rate after induction | immediately after induction
  heart rate after induction
heart rate in procedure | in procedure
  heart rate in procedure
heart rate when transited into PACU | immediately after transited into PACU (first measured data in PACU)
  heart rate into PACU
heart rate when transited out PACU | before transited out of PACU (last measured data in PACU)
  heart rate out PACU
heart rate spontaneous respiratory | immediately after recovering spontaneous respiratory
  heart rate when spontaneous respiratory recovers
heart rate effective spontaneous respiratory | immediately after effective spontaneous respiratory recovers
  heart rate when effective spontaneous respiratory recovers
heart rate LMA removal | immediately after LMA removed
  heart rate when LMA removed
baseline mean blood pressure | before induction
  mean blood pressure before induction
mean blood pressure after induction | immediately after induction
  mean blood pressure after induction
mean blood pressure in procedure | in procedure
  mean blood pressure in procedure
mean blood pressure when transited into PACU | immediately after transited into PACU (first measured data in PACU)
  mean blood pressure into PACU
mean blood pressure when transited out PACU | before transited out of PACU (last measured data in PACU)
  mean blood pressure out PACU
mean blood pressure spontaneous respiratory | immediately after recovering spontaneous respiratory
  mean blood pressure when spontaneous respiratory recovers
mean blood pressure spontaneous respiratory | immediately after effective spontaneous respiratory recovers
  mean blood pressure when effective spontaneous respiratory recovers
mean blood pressure LMA removal | immediately after LMA removed
  mean blood pressure when effective spontaneous respiratory recovers
time length of LMA removal | from the time point of the child be transited into PACU until the time point of the LMA be removed
  time length from the child transited into PACU to LMA removal
dwell time length in PACU | from the time point of the child be transited into PACU until the time point of the child be transited out of PACU
  time length of the child staying in PACU
cough | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  cough count and severity
desaturation | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  desaturation count and severity
clenching | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  clenching during LMA removal
gross body movement | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  gross body movement during LMA removal
breath holding | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  breath holding during LMA removal
airway obstruction | from the time point of the LMA be removed until the time point of the child be transited out of PACU
  airway obstruction

SECONDARY OUTCOMES:
parents' satisfaction score | up to 3 days after surgery
  questionnaire scored from 1-5 to assess the parents' satisfaction : score 1 for worst satisfied, score 5 for best satisfied
sleep quality score | up to 3 days after surgery
  questionnaire scored from 1-5 to assess the children's sleep quality : score 1 for worst sleep quality, score 5 for best sleep quality
FLACC(face,legs,activity,cry,consolability) scale score | up to 3 days after surgery
  FLACC scale scored from 0-10 to assess the children's pain after surgery: score 0 for no pain, score 10 for worst pain
anxiety score | up to 3 days after surgery
  questionnaire scored from 1-5 to assess the parents' anxiety : score 1 for no anxiety, score 5 for worst anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Wenxian Li, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and EENT hospital of Fudan University, Shanghai, Shanghai Municipality, China